CLINICAL TRIAL: NCT06782035
Title: The Influence of Periodontal Dressings (Ora-Aid) and Various Materials on the Donor Site's Quality of Life After Free Gingival Graft Surgery
Brief Title: The Effect of Periodontal Dressings and Various Materials on the Donor Site's Quality of Life After Free Gingival Graft Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Sare Eröz, Research Assistant, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-61749811-000-3341706
Record Dates: First submitted 2025-01-10; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Recession, Gingival
Keywords: Free gingival graft; Mucogingival surgery; Periodontal dressing
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: After free gingival graft surgery, different materials were applied to aid healing due to the discomfort and pain caused by the wound in the palatal donor site during the postoperative healing process. A total of 36 patients were included in the study and divided into three groups based on the material applied. The test group consisted of "Ora-Aid," while the control groups included L-PRF and the palatal stent group, with 12 patients in each group.In our study, the OHIP-14 questionnaire was used to evaluate patient satisfaction on postoperative days 3, 7, and 14. To measure pain levels on postoperative days 3, 7, and 14, the Visual Analog Scale (VAS) test was used. For VAS scoring, patients were asked to mark an integer value between 0 and 10. Wound epithelialization was assessed on days 7, 14, and 1 month postoperatively as either "present" or "absent."
Who Masked: Outcomes Assessor
Masking Description: The person assessing epithelialization does not know the group distribution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Ora-Aid (Experimental): For the test group, Ora-Aid® measuring 25 mm x 15 mm is used. After achieving hemostasis and irrigating the wound area on the palate with sterile saline, Ora-Aid® is cut to appropriate dimensions to fully cover the wound site. Using tweezers, it is separated from its transparent film layer and applied to the wound. Gentle pressure is applied for 5-10 seconds until the dressing adheres to the wound site. To enhance the stabilization of Ora-Aid® in the area, it is secured using 4/0 silk sutures with a cross-suture technique.
  Interventions: Device: Ora-Aid-Oral Wound Dressing
- L-PRF (Active Comparator): For the L-PRF group, venous blood is collected from patients using a disposable sterile syringe and placed into glass tubes without anticoagulants. The blood samples are centrifuged at 2700 rpm for 12 minutes in a centrifuge device. After the centrifugation process is completed, the clot formed in the middle layer of the tube is removed using tweezers and placed between two sterile metal plates to be compressed into a membrane. The dimensions of the obtained L-PRF membrane are adjusted according to the size of the donor site. The wound area on the palate is sutured crosswise using 4/0 silk suture material, and the L-PRF membrane is placed on the wound surface.
  Interventions: Biological: Platelet rich fibrin
- Palatal Stent (Active Comparator): For the palatal stent group, impressions are taken from patients preoperatively, and a plate is prepared. The fit of the plate is checked in the oral cavity. After the free gingival graft is harvested, hemostasis is achieved at the wound site, and the palatal stent is placed on the maxilla.
  Interventions: Device: Palatal Stent

INTERVENTIONS:
Device: Ora-Aid-Oral Wound Dressing — Intended as a physical barrier for temporary protection of oral mucosal tissue and to provide pain relief. This product is a non-eugenol protective material applied to intraoral wounds. Ora-Aid is a new concept of pasting intra-oral patch to protect the affected area such as post implant, extraction, orthodontic, and ulcers. This new concept of pasting intra-oral wound dressing is designed to protect the affected area and aid natural healing.
  Arms: Ora-Aid
Biological: Platelet rich fibrin — It has been reported that the use of Platelet-Rich Fibrin (PRF) to cover palatal wounds accelerates healing and reduces postoperative morbidity. Studies have demonstrated that PRF supports key processes in wound healing, such as "immunity," "angiogenesis," and "cellular proliferation." Its use has garnered significant interest, particularly in non-healing wounds and areas left to heal by secondary intention after surgery. Leukocyte and Platelet-Rich Fibrin (L-PRF) is frequently used in periodontal surgical applications. The platelets and growth factors it contains accelerate the healing process and facilitate tissue repair.
  Arms: L-PRF
Device: Palatal Stent — Palatal stents help prevent complications such as infection or excessive discomfort. These plates are typically customized to fit the patient's palate by taking impressions before the surgery. Once placed, they serve as a barrier, especially during the early stages of healing. Additionally, they may reduce the need for postoperative interventions, such as the use of strong painkillers.
  Arms: Palatal Stent

SUMMARY:
The inadequate width of attached gingiva, resulting from the loss of the attached gingiva band, is one of the primary mucogingival issues. Free gingival graft (FGG) is a mucogingival surgical technique used to increase the amount of attached gingiva, cover exposed root surfaces in localized gingival recessions, deepen the vestibule, and eliminate frenulum and muscle attachments. The harvested tissue is keratinized attached gingiva. Due to ease of access, the palate is most commonly preferred as the donor site.

Complications that may arise following FGG surgery are generally donor site-related. Reported complications include postoperative bleeding, recurrent herpetic lesions, delayed healing, paresthesia, mucocele, arteriovenous shunt, and postoperative pain. To aid healing and reduce discomfort and pain associated with the wound site in the palate after surgery, various materials have been applied to the donor site to facilitate recovery.

Following FGG surgery, patients will be divided into three groups based on the application of different materials to the wound site in the palate: leukocyte- and platelet-rich fibrin (L-PRF), Ora-Aid oral wound dressing, and a palatal surgical stent. In the Ora-Aid group, after harvesting the graft and placing it in the recipient site, the wound area will be irrigated with saline solution, and Ora-Aid will be trimmed to the appropriate size and shape. It will be gently pressed onto the wound for 5-10 seconds until it adheres. Ora-Aid and L-PRF will be secured to the wound site with a 4/0 silk cross suture. The Ora-Aid application will serve as the test group, the L-PRF application as the positive control group, and the palatal surgical stent as the negative control group. Randomization will be performed using a computer program.

Postoperatively, patients' pain levels will be assessed on the 3rd, 7th, and 14th days using the Visual Analog Scale (VAS) test and the OHIP-14 questionnaire. Wound site epithelialization will be evaluated during follow-up sessions on the 7th and 14th days and at 1 month. After evaluating all questionnaire results, statistical analyses will be conducted.

DETAILED DESCRIPTION:
Clinically, the gingiva is part of the oral mucosa and periodontium that covers the alveolar processes of the jaws and surrounds the cervical portions of the teeth. Topographically, it is divided into free, attached, and interdental gingiva. Following tooth eruption, the gingival margin is located 0.5-2 mm coronally to the cementoenamel junction (CEJ). Histologically, the gingiva consists of epithelium and connective tissue. Anatomically and clinically, it is divided into three distinct regions: free gingiva, interdental gingiva, and attached gingiva.

Mucogingival issues arise as a result of insufficient attached gingiva. A thick keratinized attached gingiva is necessary to protect against masticatory trauma. When attached gingiva is reduced, plaque control becomes difficult, and the area becomes prone to inflammation. For periodontal health, 2 mm of attached gingiva is considered essential. The protective barrier function of attached gingiva prevents free gingival margin movement caused by the effects of perioral muscles in cases of insufficient attached gingiva. Movement of the gingival margin increases the risk of inflammation progression and gingival recession.

Free gingival graft (FGG) is one of the mucogingival surgical procedures used to increase the amount of attached gingiva, cover exposed root surfaces in localized gingival recession, deepen the vestibule, and eliminate frenulum and muscle attachments. The harvested tissue is keratinized attached gingiva. During the FGG procedure, vestibular depth increases, allowing patients to perform brushing more comfortably. The tuberosity region, edentulous alveolar crest, and hard palate are commonly preferred as donor sites due to ease of access.

Post-FGG complications are generally related to the donor site and include postoperative bleeding, recurrent herpetic lesions, delayed healing, paresthesia, mucocele, arteriovenous shunt, and postoperative pain. The palatal donor site often causes more discomfort and pain during the healing process. To support healing, various procedures have been implemented for the palatal donor site, including palatal stent + periodontal dressing application, suturing of hemostatic sponges, and surgical cauterization or laser application.

Recent studies report that Platelet-Rich Fibrin (PRF) accelerates healing and reduces postoperative morbidity when used to cover palatal wounds. Studies have shown that PRF supports "immunity," "angiogenesis," and "cellular proliferation," which play key roles in wound healing. Its use in non-healing wounds and surgical areas left for secondary healing has garnered significant attention. Choukroun developed a method to obtain leukocyte- and platelet-rich fibrin (L-PRF) by centrifuging 9 ml of whole venous blood in non-anticoagulant tubes at 2700 rpm for 12 minutes at room temperature. The process produces three layers within the tube: platelet-poor plasma at the top, red blood cells at the bottom, and L-PRF, a fibrin structure rich in platelets and growth factors, in the middle. The L-PRF layer is extracted with forceps, separated from the red blood cell layer using scissors, and compressed between two metal trays in a sterile container to form a 1-mm-thick membrane for clinical use.

Ora-Aid wound dressing is a relatively new material used for palatal donor site healing following FGG surgery. The adhesive side of Ora-Aid is applied directly to the oral mucosa, forming a protective layer. Ora-Aid offers advantages such as aiding hemostasis, providing physical protection against food particles, bacterial irritants, and smoking, and reducing oral malodor with its natural mint flavor. Another advantage is that it naturally detaches without requiring an additional appointment for removal. Ora-Aid consists of hydrophilic high-density polymers encapsulated within water-insoluble mucoadhesive synthetic cellulose and contains vitamin E, which has wound-healing and hemostatic effects. It is available in two sizes: 50 mm × 20 mm and 25 mm × 15 mm.

After harvesting the FGG, the palatal wound is irrigated with saline solution, and Ora-Aid is trimmed to the appropriate size and shape. It is then peeled from its transparent film and applied to the wound using forceps. The dressing is gently pressed for 5-10 seconds until it adheres to the wound. Ora-Aid use has demonstrated superior results for both patients and clinicians, being effective in reducing postoperative pain and enhancing wound healing. It holds significant potential as a palatal wound dressing material.

The aim of this study is to evaluate the quality of life in patients receiving L-PRF and periodontal dressings on the donor site after free gingival graft surgery.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy Non-smoker Insufficient attached gingiva Not using any medication regularly Age 18-85 years No previous graft taken from the same area Not in pregnancy or lactation period Agreement to participate in the study and sign the "Informed Consent Form"

Exclusion Criteria:

Systemic disease Regular systemic medication use Under 18 years old Pregnant or breastfeeding women Smoker Previous graft taken from the same area

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
"Patient Satisfaction Data Assessed with the Oral Health Impact Profile-14 (OHIP-14) Questionnaire" | Postoperative days 3, 7, and 14
  In our study, the OHIP-14 questionnaire was used to evaluate patient satisfaction on postoperative days 3, 7, and 14. The OHIP-14 questionnaire comprises 14 questions (S1-S14) related to functional limitation (S1-S2), physical pain (S3-S4), psychological discomfort (S5-S6), physical disability (S7-S8), psychological disability (S9-S10), social disability (S11-S12), and handicap (S13-S14). Each question was scored on a 5-point Likert scale.
Use of Visual Analog Scale (VAS) for Pain Measurements | Postoperative days 3, 7, and 14
  The Visual Analog Scale (VAS) test is used to measure pain levels in patients on postoperative days 3, 7, and 14. For VAS scoring, patients are asked to mark an integer value between 0 and 10.

SECONDARY OUTCOMES:
Hydrogen Peroxide Test for the Presence of Epithelialization | Postoperative day 7, day 14, and month 1.
  Wound epithelialization is assessed on days 7, 14, and 1 month as "present/absent."

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University Faculty of Dentistry Department of Periodontology, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No